CLINICAL TRIAL: NCT05059106
Title: EFFECTIVENESS, SAFETY AND IMMUNOGENICITY OF THE HALF DOSE OF THE VACCINE ChadOx1 nCoV-19 (AZD1222) for COVID-19
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Federal University of Espirito Santo (Other)
Collaborators: Centro de Pesquisas René Rachou (Other Government); Escola Nacional de Saúde Pública Sérgio Arouca/Fiocruz (Unknown); Oswaldo Cruz Foundation (Other); Escola Superior de Ciências da Santa Casa de Misericórdia de Vitória (Unknown)
Responsible Party: Principal Investigator, Valéria Valim, Professor, Federal University of Espirito Santo
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: FUES02
Record Dates: First submitted 2021-09-24; First posted 2021-09-28 (Actual); Last update posted 2021-09-28 (Actual); Status verified 2021-09

CONDITIONS: SARS-CoV-2
Keywords: vaccines; immunity; covid-19
MeSH Terms: conditions — COVID-19 | interventions — ChAdOx1 nCoV-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Experimental): Half dose of ChAdOx1 nCoV-19 (AZD1222) ) in a 2-dose schedule with an interval of 8 weeks.
  Interventions: Biological: Half dose of ChAdOx1 nCoV-19 (AZD1222)
- Group 2 (Active Comparator): Standad dose of ChAdOx1 nCoV-19 (AZD1222) in a 2-dose schedule with an interval of 8 weeks.
  Interventions: Biological: Standard dose of ChAdOx1 nCoV-19 (AZD1222)

INTERVENTIONS:
Biological: Half dose of ChAdOx1 nCoV-19 (AZD1222) — Vaccination with reduced dose (half dose) of ChAdOx1 nCoV-19 (AZD1222), in a 2-dose schedule with an interval of 8 weeks, including all adults aged 18 to 49 years, from non-priority groups, from Viana city - Espírito Santo (ES)/Brazil.
  Arms: Group 1
Biological: Standard dose of ChAdOx1 nCoV-19 (AZD1222) — Vaccination with standad dose of ChAdOx1 nCoV-19 (AZD1222), in a 2-dose schedule with an interval of 8 weeks, in external cohort of health workers aged 18 to 49 years.
  Arms: Group 2

SUMMARY:
This study is clinical trial (intervention study with external comparison group) to test vaccination with reduced dose (half dose) of ChAdOx1 nCoV-19 (AZD1222), in a 2-dose schedule with an interval of 8 weeks, including all adults aged 18 to 49 years from Viana city - Espírito Santo (ES)/Brazil, on the incidence of new cases over 12 months following treatment, compared to an external group from same state and adjusted for socio-demographic and epidemiological variables.

DETAILED DESCRIPTION:
This study is clinical trial (intervention study with external comparison group) to test vaccination with reduced dose (half dose) of ChAdOx1 nCoV-19 (AZD1222), in a 2-dose schedule with an interval of 8 weeks, including all adults aged 18 to 49 years from Viana city - Espírito Santo (ES)/Brazil, on the incidence of new cases over 12 months following treatment, compared to an external group from same state and adjusted for socio-demographic and epidemiological variables. Cellular and humoral immunity will be studied in a representative sub-sample compared to an external reference group (cohort of health workers) vaccinated with standard dose. The outcomes will be evaluated at 28 days after the second dose and follow-up after 6 months and 12 months. The main outcome will be to decrease in 60% the incidence of new cases over 6 months after receiving the vaccine. The clinical epidemiological variables will be obtained from e-SUS VS, e-SUS notifica and datasus: number of cases, number of deaths with specific ICD for covid-19, number of hospital admissions for covid-19; number of ICU admissions for the treatment of SARS, total number of tests (RT-PCR) performed and positive. The cellular and humoral immune response will be assessed by viral neutralization assay (neutralizing antibody test), serological assay by chemiluminescence, determination of specific IgM and IgG profiles, measurement of systemic soluble factors (chemokines, cytokines and growth factors), stimulation antigen-specific peripheral blood mononuclear cells in vitro and investigation of memory T and B lymphocytes and intracytoplasmic cytokines. It is estimated to include 29,637 people in the study, to reach 85% vaccination cover of individuals aged 18-49 years. The subsample size immunogenicity test is 600 individuals from the eligible population, estimating losses of 15% and study power of 90%, alpha error of 1%. The hypothesis of the study is that the reduction in the incidence of covid-19 and the cellular and humoral immune response achieved with a half dose will be similar to the reduction expected with the standard dose.

ELIGIBILITY:
Inclusion Criteria:

- residents of Viana, Espírito Santo, aged between 18 and 49 years

Exclusion Criteria:

* Pregnant women;
* History of severe allergic reaction (anaphylaxis) to any previously administered vaccine;
* Having received another vaccine in the last 14 days;
* Belonging to a priority risk group for vaccination, as per the PNI recommendations;
* Have fever or flu-like symptoms;
* Have previously received any vaccine for covid-19 at any time;
* Recent diagnosis of covid-19 with onset of symptoms 28 days before vaccination;
* Disorders of coagulation and use of anticoagulants.

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 29637 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2022-06-01 (Estimated); Study Completion 2022-10-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of new cases | 12 months
  Incidence of new cases over 12 months following treatment

SECONDARY OUTCOMES:
Number of deaths | 12 months
  Number of deaths with specific ICD for covid-19
number of hospital admissions | 12 months
  number of hospital admissions for covid-19
number of intensive care unit (ICU) admissions | 12 months
  number of intensive care unit (ICU) admissions for the treatment of SARS
number of tests (RT-PCR) | 12 months
  number of tests (RT-PCR) performed and positive
Viral Neutralization Assay | 4 and 8 months
  Neutralizing antibody titers will be expressed by the ability of antibodies to neutralize up to 50% the number of plaques (PRNT50). Title > 1:50 will be considered positive.
serological assay | 8 and 10 months
  Serological test by chemiluminescence. Results are expressed in U/mL and data interpretation will be done as follows: <0.8 U/mL = non-reactive sample; ≥0.8 U/mL = reactive sample.
IgM | 8 and 10 months
  Determination of specific IgM profile. Results will be expressed in fluorescence intensity or pg/ml.
IgG | 8 and 10 months
  Determination of specific IgG profile. Results will be expressed in fluorescence intensity or pg/ml.
systemic soluble factors | 8 and 10 months
  Dosage of soluble systemic factors (chemokines, cytokines and growth factors). Results will be expressed in pg/ml.
Antigen-specific stimulation of peripheral blood mononuclear cells | 10 and 12 months
  Antigen-specific stimulation of peripheral blood mononuclear cells in vitro. The results will be expressed in percentage positive frequency for a specific cell phenotype.
Lymphocyte investigation | 10 and 12 months
  Investigation of memory T and B lymphocytes. The results will be expressed in percentage positive frequency for a specific cell phenotype.
Cytokine investigation | 10 and 12 months
  Investigation of intracytoplasmic cytokines. The results will be expressed in percentage positive frequency for a specific cell phenotype.

OTHER OUTCOMES:
Adverse events | 14 months
  All adverse events will be followed up to establish severity and causal correlation. There will be surveillance of deaths and will be reported to the ethics committee.

CONTACTS AND LOCATIONS:
Locations (1):
- Federal University of Espirito Santo, Vitória, Espírito Santo, Brazil

REFERENCES:
- [Derived] Medeiros-Junior NF, Gouvea MDPG, Camacho LAB, Villela DAM, Lima SMB, Schwarcz WD, Azevedo AS, Neto LFP, Domingues CMAS, Fantoni RNDS, Forechi L, Ruchdeschel T, Albertino LF, Pereira M, Rizzi RB, Muniz SM, Santos HCD, de Oliveira Roza TL, Oliveira YGP, Dias LH, Miyamoto ST, Tapia KRL, Lyra DGP, Jubini JD, Burian APN, Moulaz IR, Araujo MF, Tort LFL, Oliveira ACA, Oliveira Prado R, Pereira AAS, Miranda VHS, Speziali E, Costa-Pereira C, Alves CC, Carvalho KRA, Dos Santos LM, Oliveira-Carvalho N, Oliveira G, Santos TMAFD, Figueiredo ACC, Costa-Rocha IA, Campi-Azevedo AC, Peruhype-Magalhaes V, Garcia CC, Siqueira MM, Antonelli LRDV, Coelho-Dos-Reis JGA, Teixeira-Carvalho A, Mill JG, Martins-Filho OA, Valim V. Third Booster Half Dose of ChAdOx1-nCov-19 Is Effective, Safe, and Induces Long-Duration Humoral and Cellular Immune Response to Omicron: 1-Year Follow-Up of Viana Study. Vaccines (Basel). 2025 Oct 30;13(11):1113. doi: 10.3390/vaccines13111113. PMID 41295486